CLINICAL TRIAL: NCT00174538
Title: The Effects of Cytochrome P450 2D6 Genotype on Pain Management With Codeine in Sickle Cell Disease
Brief Title: Codeine in Sickle Cell Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR007111; FEN-EMR-4007
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2005-07

CONDITIONS: Sickle Cell Disease
Keywords: codeine; pain; CYP2D6; genotype; morphine; sickle cell; pharmacokinetic
MeSH Terms: conditions — Anemia, Sickle Cell; Pain | interventions — Codeine

INTERVENTIONS:
Drug: Codeine (30 mg)

SUMMARY:
The objective of this study is to determine if a subject's genetic make-up would affect the treatment response to codeine in subjects with sickle cell disease.

DETAILED DESCRIPTION:
People with sickle cell disease require oral pain medications to manage an acute pain crisis. Sometimes these individuals fail to obtain adequate pain relief with the medications prescribed for outpatient use resulting in emergency room visits and hospital admissions. Subsequently, many patients are admitted to the hospital for pain management for a few days until the pain crisis resolves. The most common medications prescribed to sickle cell individuals for outpatient use include codeine and hydrocodone containing medications (i.e. Tylenol #3™, Vicodin™, Lortab™). These medications must be broken down in the body to make the active pain reliever (morphine or hydromorphone, respectively). Some individuals may not be able to break down these medications to the active pain reliever; therefore, these individuals will likely continue to experience pain unless they take other pain medications. We will determine whether genotype estimates the ability of CYP2D6 to break down codeine to the active pain reliever in individuals with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Sickle cell disease (HbSS)
* Hydrocodone- or codeine-containing medications to manage an acute pain crisis in the past

Exclusion Criteria:

* Renal dysfunction, serum creatinine (SCr) > 2.0 mg/dl
* Hepatic dysfunction, AST, ALT or direct bilirubin > 3 x upper limit of normal (ULN)
* Codeine allergy
* Medications shown to induce or inhibit CYP2D6
* Women who are pregnant or breast feeding
* Unable to provide written, informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-03; Study Completion 2005-12

PRIMARY OUTCOMES:
Plasma morphine and codeine concentrations
CYP2D6 genotype

SECONDARY OUTCOMES:
Disease severity
Hospitalizations and admissions

CONTACTS AND LOCATIONS:
Overall Officials: Stacy S. Shord, PharmD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Medical Center, Chicago, Illinois, United States